CLINICAL TRIAL: NCT04817657
Title: COVID Vaccine VAC31518 Pre-approval Access Study
Brief Title: Pre-approval Access for Janssen's COVID Vaccine VAC31518 for Treating Physician Use
Status: No longer available | Type: Expanded Access
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR109001; VAC31518COV4006 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2021-03-24; First posted 2021-03-26 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Healthy
MeSH Terms: interventions — Ad26COVS1

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Biological: Ad26.COV2.S — Participants will be administered 0.5 milliliter suspension of Ad26.COV2.S 1*10^11 virus particles per milliliter (vp/ml) as intramuscular injection.
  Other Names: VAC31518, JNJ-78436735

SUMMARY:
The purpose of this Pre-approval access (PAA) program is to provide VAC31518 (Ad26.CoV2.S) vaccine for the prevention of coronavirus disease-2019 (COVID-19) infection. This PAA program may be considered to protect participants against a serious/life-threatening diseases or conditions, where there are no alternative treatments available.

Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC